# Insights from Participants: Candid Accounts of Schizophrenia Clinical Trials Patients

An Informed Consent Form (ICF) For <u>Power Clinical Trial's</u> Schizophrenia Observational Study

Date: July 7, 2023

Understanding the Informed Consent Document

You are presented with an opportunity to participate in this observational clinical trial by filling up this form. This crucial document aims to shed light on the intricate workings of the study, encompassing its overarching objectives, the step-by-step process, and a balanced portrayal of the potential benefits and drawbacks. As you navigate this decision, it becomes paramount to engage in thoughtful deliberation and seek guidance from a trusted confidant or your care team. If any questions or uncertainties arise regarding the information provided, feel free to approach the researcher for further elucidation.

# The Purpose Behind This Clinical Trial

Schizophrenia is a mental health disorder that affects how a person thinks, feels, and behaves. It is characterized by a combination of symptoms, including hallucinations (seeing or hearing things that are not there), delusions (strongly held beliefs that are not based in reality), disorganized thinking and speech, diminished emotional expression, and difficulties in social interaction and functioning.

The primary objective of conducting clinical trials for schizophrenia is to evaluate the safety and efficacy of emerging treatments. Through these trials, researchers strive to determine the superiority of new treatments over existing ones, thereby gathering compelling evidence to endorse their utilization within the general populace.

This study seeks to delve into the firsthand experiences of patients diagnosed with schizophrenia who partake in a separate clinical trial featuring a specific medical intervention. The primary emphasis will be on meticulously tracking the rates of trial completion and withdrawal among these individuals.

The Significance of Observational Clinical Trials in Advancing Medical Knowledge

By joining this medical trial, you will be participating in an observational study, a unique type of clinical trial designed to gather essential information by closely observing individuals while maintaining their existing care plans without any modifications.

Throughout the trial, researchers will attentively observe your progress and meticulously measure the outcomes of your condition without any interventions. These trials serve as invaluable tools for gaining a profound understanding of the natural progression of a specific condition and its impact on individuals who have been diagnosed. Your active participation in this observational study will contribute significantly to the advancement of medical knowledge, leading to improvements in the care provided to individuals facing the same condition.

# Comparing Schizophrenia Clinical Trials

While the current clinical trial takes an observational approach without administering specific treatments or interventions, it is important to acknowledge the presence of other clinical trials for schizophrenia that follow an interventional path, requiring participants to undergo targeted treatment regimens.

To make an informed decision about potential participation in a clinical trial, conducting thorough research and performing comparative analyses of different studies is crucial. Valuable information about <u>schizophrenia studies</u> can be obtained from clinicaltrials.gov or by visiting Power's website, which provides insights into ongoing <u>schizophrenia clinical trials</u> open for recruitment. By dedicating time and effort to understanding the various types of clinical trials available, you can confidently navigate your options and make a discerning choice regarding your suitability for trial participation.

## Participating in an Observational Clinical Trial

As a participant in this observational clinical trial, we greatly appreciate your contribution and seek to gather valuable insights into your experiences. This will be achieved through the completion of questionnaires every two weeks, which will require approximately 20-30 minutes of your time. Additionally, periodic check-in calls will be conducted on a quarterly basis for the duration of your participation in the trial.

It is important to emphasize that your participation in the survey component of this trial is entirely voluntary. You have the autonomy to choose which questions to answer, and at any point, you may decide to discontinue your involvement. We understand that the decision to participate in a clinical trial is personal, and we are dedicated to providing support throughout your journey. Your privacy and comfort are of the utmost importance, and we will fully respect your decision-making process throughout the trial.

#### Ensuring Anonymity in Survey Responses

Protecting the privacy of your information is our top priority in this clinical trial. To ensure complete anonymity, we kindly ask you to avoid including any personal or identifying details in your questionnaire responses. The research team will take all necessary precautions to safeguard your confidentiality. However, it is important to acknowledge that specific legal obligations may require the disclosure of your data in certain situations.

## Advancing Schizophrenia Research Opportunities

While immediate benefits may not be readily noticeable for participants in this observational clinical trial, their involvement can have a far-reaching impact on the lives of others. The data collected from participants will play a vital role in enhancing the enrollment process for future individuals with schizophrenia, making it easier for them to access valuable medical research opportunities. By joining this clinical trial, individuals have a distinctive opportunity to contribute to the improvement of future schizophrenia patients' well-being and actively contribute to the advancement of medical research.

## Mitigating Risks in Observational Trials

Clinical trials play a crucial role in advancing medical knowledge but may involve potential health risks, especially when new treatments are being evaluated. However, it is important to highlight that our observational clinical trial eliminates such risks, as participants are not exposed to any new interventions. Instead, they are closely observed, and outcomes are measured to ensure their safety throughout the duration of the trial.

The protection of participant confidentiality is of utmost importance in clinical trials, and our medical study employs robust measures to ensure the privacy of participant information. All data collected from participants is anonymized, and access to this information is strictly limited to the research team.

Furthermore, comprehensive security protocols are implemented to safeguard all records, including call logs, online transactions, forms, and surveys. These records are securely stored using encryption and password protection, guaranteeing the confidentiality and protection of participant information. This rigorous approach ensures that participant data remains confidential and shielded from unauthorized access, prioritizing the privacy and trust of all individuals involved in the trial.

## **Understanding Patients' Decision-Making**

We cordially invite you to voluntarily participate in an observational research study aimed at exploring the factors that drive patients' decisions to take part in clinical trials for schizophrenia. It is essential to emphasize that this study does not involve proposing new treatment protocols or making any modifications to your current treatment plan.

Throughout this study, the researcher will conduct interviews to gather valuable information about your experiences. However, aside from the interviews, all aspects of your treatment and care will remain unchanged. The researcher will neither provide a diagnosis nor recommend any specific course of treatment. The primary objective of this study is to collect data for research purposes.

To be eligible for participation, it is necessary for you to be currently enrolled in another clinical trial for schizophrenia. By delving into the motivations behind your decision to participate and the factors influencing your determination to continue or discontinue treatment in that trial, we aim to gain deeper insights into patients' perspectives and experiences within clinical trials for schizophrenia.

Please remember that your participation in this study is entirely voluntary, and you have the freedom to withdraw at any time if you feel uncomfortable. Your decision to withdraw will not impact any of your legal rights, and your ongoing treatment plan in the other clinical trial will remain unaffected.

#### Resources for Informed Engagement in Clinical Trials

For those seeking a deeper understanding of representation in clinical trials, there is a wealth of online resources available to explore this crucial topic. These resources offer valuable insights into the challenges and opportunities surrounding diversity in clinical research, providing a comprehensive perspective:

Kim, Janice, Robert Kester, and Gideon Blumenthal. "Clinical trial diversity in oncology: FDA takes action with post—marketing requirements or commitments." *The Oncologist* 27, no. 12 (2022): 993-997.

MacLennan, Demi L., Jennifer L. Plahovinsak, Rob J. MacLennan, and Carolynn T. Jones. "Clinical trial site perspectives and practices on study participant diversity and inclusion." *Clinical Pharmacology & Therapeutics* 113, no. 3 (2023): 670-679.

By engaging with these resources, individuals can gain valuable knowledge to inform their own involvement in clinical trials and actively contribute to promoting diversity and inclusivity in the field of medical research.

# Acknowledging Informed Consent

I hereby confirm that I have taken sufficient time to thoroughly read and comprehend the contents of the informed consent form, either independently or with the assistance of a trusted individual who has read it to me. All of my questions and concerns have been adequately addressed to my complete satisfaction.

I am fully aware that my participation in this study is entirely voluntary, and I have the right to withdraw my consent at any time, without the need to provide a reason or face any financial obligations. I have been informed that I will receive a copy of this informed consent form for my personal records.

| After careful consideration and thoughtful reflecti<br>willingly give my consent to participate in this stu | • |
|---|---|
| Printed Name of Participant | |
| Participant Signature | |
| Date | |
| Confirming Informed Consent | |
| I hereby confirm that I have diligently reviewed the participant, ensuring their comprehensive understand potential risks and benefits, and other essential actinical trial. | standing of the purpose, methodologies, |
| During the discussion, I fostered a conducive ento ask questions and seek clarifications, effective misconceptions they may have had. It is crucial to participation in this trial is entirely voluntary, grantheir consent at any point without facing any final | ely addressing any concerns or o emphasize that the participant's ting them the autonomy to withdraw |
| Following their expression of consent, a copy of participant for their personal reference. | this document was provided to the |
| Printed Name of Person Taking Consent | |
| Signature of Person Taking Consent | |
| Date | |